CLINICAL TRIAL: NCT02270788
Title: A Phase I Pharmacokinetic, Pharmacodynamic and Feasibility Study of Crenolanib in Combination With Sorafenib in Patients With Refractory or Relapsed Hematologic Malignancies (ARO-008)
Brief Title: Crenolanib in Combination With Sorafenib in Patients With Refractory or Relapsed Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Arog Pharmaceuticals, Inc. (Industry); Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELHEM2; NCI-2014-01784 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — crenolanib; Sorafenib; Methotrexate; Hydrocortisone; Cytarabine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): All participants who consent and are enrolled on the study.
  Interventions: Crenolanib, sorafenib, triple intrathecal chemotherapy (methotrexate, hydrocortisone and cytarabine with leucovorin).
  Interventions: Drug: Crenolanib; Drug: Sorafenib; Drug: methotrexate, hydrocortisone and cytarabine with leucovorin

INTERVENTIONS:
Drug: Crenolanib — Day 1 of Course 1: once followed by pharmacokinetic analysis. Days 2-28 of cycle 1: 3 times per day Crenolanib dose will not be adjusted unless the participant experiences side effects.
  All subsequent courses: 3 times per day on Days 1-28. At least 50% of participants in each dose level must be ≤ 18 years old.
  Other Names: CP-868,596; IND 112201
Drug: Sorafenib — Days 8-28 of course 1: given orally once each day.
  All subsequent courses: given orally on days 1-28 once per day
  This is a dose-finding study for the use of sorafenib in combination with crenolanib. Different doses will be given to several participants, with the first participants receiving a lower dose than typically used in children as a single agent. If the drug does not cause serious side effects, it will be given to other study participants at a higher dose. If side effects occur, the dose will be lowered.
  Other Names: Sorafenib tosylate; BAY-43-9006; Nexavar®
Drug: methotrexate, hydrocortisone and cytarabine with leucovorin — Triple IT therapy includes methotrexate, hydrocortisone and cytarabine with leucovorin rescue given on day 8. All participants will receive one IT chemotherapy on Day 8 of the first cycle. If they do not have leukemia cells in their spinal fluid, they will receive only one IT chemotherapy per cycle. If leukemia cells are present in their spinal fluid, they will receive IT chemotherapy weekly during the course. Triple IT therapy will be repeated on Day 1 of Cycle 2 and with each subsequent cycle in all participants.
  Other Names: Triple IT chemotherapy

SUMMARY:
PRIMARY OBJECTIVE:

This is a pilot study to characterize the toxicity profile, to determine the maximum tolerated dose of the combination of crenolanib and sorafenib, and to determine the feasibility of administering these drugs in patients with relapsed or refractory hematologic malignancies, including acute myeloid leukemia (AML), AML with prior myelodysplastic syndrome (MDS), and myeloperoxidase (MPO)-positive mixed phenotype acute leukemia with FLT3-internal tandem duplication (ITD) and tyrosine kinase domain (TKD) mutations.

The study will include two phases:

* The dose-escalation phase will characterize the dose-limiting toxicities (DLTs) and determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of crenolanib when given in combination with sorafenib.
* The dose-expansion cohort will further assess the safety and explore the efficacy of this combination.

DETAILED DESCRIPTION:
Each course of therapy will be 28 days (±5 days), unless disease progression is seen while on the combination of crenolanib with sorafenib. Patients may receive subsequent courses (up to a total of 365 days) if there is no disease progression or unacceptable toxicity.

In Day 1 of Course 1, crenolanib is given once in the morning followed by characterization of the pharmacokinetic profile over the following 24-hour period. Starting with day 2 of Course 1, crenolanib will be given 3 times per day through day 28. On Days 8 to 28 of Course 1, sorafenib will be given once per day. Inter-patient dose escalation or de-escalation of crenolanib will be performed based on tolerability and toxicity.

Response will be assessed on days 8 and at end of course. If disease progresses prior to day 8, then sorafenib can be given before day 8.

In subsequent courses (up to 365 days), crenolanib and sorafenib are given on days 1 through 28. The treating physician may increase or decrease the sorafenib dose and frequency of administration per the trial's dosing table on the basis of effects and tolerability. If necessary, the crenolanib dose can be decreased per protocol.

Maintenance therapy must start no sooner than 30 days and no later than 120 days after hematopoietic stem cell therapy (HSCT). Single agent crenolanib will start at the last dose tolerated prior to HSCT. Crenolanib maintenance can be given for up to 365 days and additional therapy can be provided after discussion after discussion with the PI, in patients who continue to benefit after 1 year.

ELIGIBILITY:
Inclusion Criteria - Initial Enrollment:

* Participant has a relapsed or refractory hematologic malignancy (with any measurable disease) with FLT3-ITD or TKD mutations and one of the following diagnoses:

  * Acute myeloid leukemia (AML)
  * AML with prior myelodysplastic syndrome (MDS)
  * Myeloperoxidase (MPO)-positive mixed phenotype acute leukemia
* Participant's disease has relapsed after, is refractory to induction and/or salvage therapy, or has relapsed after hematopoietic stem cell transplant (HSCT).
* Participant disease tested positive for FLT3-ITD or -TKD within 60-day screening period.
* Participant's age is 1 to 25 years, inclusive (St. Jude participants must be aged 1 to 25 years, inclusive).
* Karnofsky or Lansky performance score is > 60%. The Lansky performance score should be used for participants < 16 years and the Karnofsky performance score for participants ≥ 16 years.
* Adequate organ function defined as:

  * Bilirubin ≤1.5 x upper limit of normal (ULN)
  * ALT ≤ 3 x ULN and AST ≤ 3 x ULN
  * Serum creatinine ≤1.5 x ULN
* Participant must have recovered from the acute side effects of all prior anti-cancer therapy, and:

  * At least 2 weeks have elapsed since prior systemic cytotoxic chemotherapy (except intrathecal chemotherapy, hydroxyurea, low-dose cytarabine, and/or low dose maintenance therapy such as vincristine, mercaptopurine, methotrexate or glucocorticoids), and
  * If the participant received a prior allogeneic HSCT, at least 30 days have elapsed and there is no evidence of clinically significant graft versus host disease requiring treatment and/or have > grade 2 persistent non-hematologic toxicity related to a transplant

Exclusion Criteria - Initial Enrollment:

* Concurrent chemotherapy, or targeted anti-cancer agents, other than hydroxyurea, low-dose cytarabine, intrathecal therapy and/or low dose maintenance therapy such as vincristine, mercaptopurine, methotrexate or glucocorticoids.
* Patient with concurrent severe and/or uncontrolled medical conditions that, in the opinion of the investigator, may impair participation in the study or the evaluation of safety and/or efficacy.
* Known HIV infection or active hepatitis B (defined as hepatitis B surface antigen-positive) or C (defined as hepatitis C antibody-positive).
* Prior crenolanib treatment for a non-leukemic indication.
* Major surgical procedures within 14 days of Day 1 administration of crenolanib.
* Pregnant or lactating (female participant of childbearing potential must have negative serum or urine pregnancy test required within 7 days prior to start of treatment).
* Male or female participant of reproductive potential must agree to use appropriate methods of contraception for the duration of study treatment and for at least 30 days after last dose of protocol treatment
* Inability or unwillingness or research participant or legal guardian/representative to give written informed consent.

Inclusion Criteria - Maintenance Therapy After HSCT:

* Patient must have received crenolanib on this protocol prior to HSCT to continue on to maintenance.
* Patient must be within 30 - 120 days after hematopoietic stem cell transplant (HSCT).
* Response to previous treatment on this protocol: at least resistant disease with clinical benefit or better response.
* Patient is off or on a stable dose of immunosuppressive drugs for management or prophylaxis of graft-versus-host-disease (GVHD) (defined as no escalation of therapy for GVHD) within 14 days prior to starting crenolanib.
* Patient must have recovered from acute side effects of HSCT, defined as having <Grade 2 non-hematological toxicity related to the transplant (exceptions are alopecia and other non-acute toxicities).
* Adequate hematopoietic recovery (ANC >500/mm^3 and platelet count >50,000/mm^3)
* Research participant or legal guardian/representative is able and willing to give written informed consent.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Through Day 28 of Course 1
  Any participant who experiences DLT at any time during cycle 1 of protocol therapy is considered evaluable for toxicity. Participants without DLT and can be followed for 28 days are also considered evaluable for toxicity. Participants who are not evaluable for toxicity (such as those removed early from therapy to start alternate therapy) at a given dose level will be replaced.
Maximum tolerated dose (MTD) | Through Day 28 of Course 1
  The MTD is empirically defined as the highest dose level at which six participants have been treated with at most one participant experiencing a DLT and the next higher dose has been determined to be too toxic. If the lowest dose level studied is too toxic or the highest dose level studied is considered safe, the MTD will not have been considered estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroto Inaba, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://stjude.org/protocols